CLINICAL TRIAL: NCT05370755
Title: A Phase Ia /Ib Dose Finding Study to Evaluate the Safety, Tolerability and Pharmacokinetics and Preliminary Anti-Tumor Activity of ICP-189 and ICP-189 in Combination With Anti-PD-1 Monoclonal Antibody in Patients With Advanced Solid Tumors
Brief Title: A Study of ICP-189 and ICP-189 in Combination With Anti-PD-1 Monoclonal Antibody in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00801
Record Dates: First submitted 2022-04-22; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Patients With Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ia: ICP-189 Dose Escalation (Experimental)
  Interventions: Drug: ICP-189

INTERVENTIONS:
Drug: ICP-189 — Administered orally

SUMMARY:
A Dose finding Study to Evaluate the Safety, Tolerability and Pharmacokinetics and Preliminary Anti-Tumor Activity of ICP-189 Tablets and ICP-189 Tablets in Combination with Anti-PD-1 Monoclonal Antibody in Patients with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
2. Patients with histologically confirmed locally advanced unresectable or metastatic solid tumors;
3. At least one measurable lesion according to RECIST 1.1.

Exclusion Criteria:

1. Patients who have had other cancer(s) within 5 years prior to the first dose, except for locally curable cancers that have been apparently cured;
2. Patients with unstable primary central nervous system (CNS) tumors or CNS metastases;
3. Patients who have an active autoimmune disease or have had an autoimmune disease with risk of recurrence;
4. Patients who have active or history of interstitial lung disease or non-infectious pneumonia;
5. Patients who have a history of severe allergic reaction to any component of ICP-189 tablets or anti-PD-1 antibody (> grade 3 assessed by CTCAE 5.0).

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse event (AE) of ICP-189 assessed by NCI-CTCAE V5.0 | through study completion, an average of 2 years
  To assess the safety and tolerability of ICP-189 in patients with advanced solid tumors.
Dose-Limiting Toxicities (DLTs) | through study completion, an average of 2 years
  Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs).
Recommended Phase 2 Dose (RP2D) and/or maximum tolerated dose (MTD) | through study completion, an average of 2 years
  To preliminarily determine the PR2D and the MTD of ICP-189 in patients with advanced solid tumors

SECONDARY OUTCOMES:
The maximum plasma concentration observed (Cmax) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-189 in patients with solid tumors.
Time of maximum observed plasma concentration (Tmax) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-189 in patients with solid tumors.
Elimination half-life (t1/2) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-189 in patients with solid tumors.
Area under plasma concentration-time curve (AUC0-t and AUC0-∞) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-189 in patients with solid tumors.
Apparent clearance (CL/F) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-189 in patients with solid tumors.
Apparent volume of distribution (Vz/F) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-189 in patients with solid tumors.
The objective response rate (ORR) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-189.
Duration of response (DoR) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-189.
Progression-free survival (PFS) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-189.
Overall survival (OS) | through study completion, an average of 3.5 years
  To evaluate the preliminary anti-tumor activity of ICP-189.

OTHER OUTCOMES:
Pharmacodynamics | through study completion, an average of 2 years
  On-treatment versus baseline comparison of PD biomarkers e.g., phosphorylated form of extracellular signal-regulated kinase (pERK), dual specificity phosphatase 6 (DUSP6).

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China